CLINICAL TRIAL: NCT01511211
Title: Effect of Dexamethasone on Duration of Analgesia After Ultrasound-Guided Femoral, Obturator, and Popliteal Blocks With Ropivacaine in Total Knee Arthroplasty
Brief Title: Duration of Leg Nerve Blocks With Dexamethasone Added to Local Anesthetic
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Other researchers have published results on a similar trial
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Nicholas Lam, Associate Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNMLAMLLDEX
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Pain; Total Knee Arthroplasty
Keywords: Dexamethasone; lower limb block; ultrasound guided femoral nerve block; ultrasound guided obturator nerve block; ultrasound guided sciatic nerve block; ropivacaine; total knee arthroplasty; Post surgical pain after total knee arthroplasty
MeSH Terms: conditions — Pain | interventions — Dexamethasone; Calcium Dobesilate; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ropivacaine + Dexamethasone Combination (Experimental)
  Interventions: Drug: Dexamethasone
- Ropivacaine-Only Block (Active Comparator)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Dexamethasone — 2 cc of 4 mg/cc dexamethasone will be added to 38 cc of 0.5% ropivacaine solution. Of this combination, 15 cc will be used for a femoral nerve block, 20 cc for the popliteal nerve block, and 5 cc for the obturator nerve block. In addition, 2 cc of normal saline will be added to the patient's IV to maintain blinding.
  Other Names: Decadron
  Arms: Ropivacaine + Dexamethasone Combination
Drug: Ropivacaine — 2 cc of normal saline will be added to 38 cc of 0.5% ropivacaine solution. Of this combination, 15 cc will be used for the femoral nerve block, 20 cc for the popliteal nerve block, and 5 cc for the obturator nerve block. In addition, 2 cc of 4 mg/cc dexamethasone will be added to the patient's IV.
  Other Names: Naropin
  Arms: Ropivacaine-Only Block

SUMMARY:
This is a Randomized Double blinded controlled trial on the effect of adding dexamethasone to Ropivacaine on the duration of pain relief for ultrasound guided femoral, obturator and popliteal block after total knee replacement surgery.

DETAILED DESCRIPTION:
This is a double blinded randomized controlled trial on the effect on duration of action when we add dexamethasone to our 3 routine peripheral nerve blocks (femoral, obturator and sciatic nerve) for total knee replacement surgery.

Technique:

A computer generated randomization will determine if dexamethasone 8mg (2 cc of 4mg/cc) will be given to the patient intravenously or mixed with the ropivacaine for the lower limb blocks. A sham 2 ml of normal saline will be given in the other route. For example, if the patient is assigned to the Ropivacaine + Dexamethasone Combination arm, 2 ml of dexamethasone will be drawn up and labeled "PNB" (peripheral nerve block) by a person not involved in the block or anesthetic management of the patient and given to the regional anesthesiologist to add to their local anesthetic solution. Another 2 ml of normal saline labeled (IV) will be drawn up by the same person and the sham will be given to the anesthesia team taking care of the patient during surgery for them to give it to the patient intravenously just before the start of the surgery.

Alternatively, if the patient is assigned to the Ropivacaine-Only Block arm, a person not involved in the patient care will draw up 2 ml of normal saline and label it "PNB" and give it to the regional anesthesiologist and 2ml of dexamethasone and label it "IV" to the anesthesia team taking care of the patient during surgery for them to give it to the patient intravenously just before the start of surgery.

Randomization:

70 patients will be randomly selected to receive either:

1. Combo A = 38 cc of 0.5% Ropivacaine with 2 cc of 4mg/cc Dexamethasone in the lower limb blocks PLUS 2cc normal saline intravenously. 15 cc of solution will be used for the femoral block, 20 cc for the popliteal block and 5 cc will be used for the obturator block.
2. Combo B = 38 cc of 0.5% Ropivacaine with 2 cc of saline in the lower limb block PLUS 2cc of 4mg/cc of Dexamethasone intravenously. 15 cc of solution will be used for the femoral block, 20 cc for the popliteal block and 5 cc will be used for the obturator block.

Blinding:

A sealed envelope will be given to an anesthesia provider not involved in the peripheral nerve block, follow up assessment of the block or provide perioperative anesthesia care to the patient. This person would draw up 2 cc of dexamethasone and 2 cc of normal saline and label them for intravenous (IV) injection or addition to the ropivacaine mixture in the lower limb block (PNB) depending on the instructions in the envelope.

The anesthesia provider performing the peripheral nerve block, providing perioperative anesthesia care including the general anesthesia or monitored anesthesia care nor the anesthesia providers assessing the patients block will not have information regarding the route of dexamethasone given.

Block performance:

All blocks are to be performed by 1 of our 7 regional anesthesiologists with expertise in ultrasound-guided lower limb blocks who will be blinded to the presence of dexamethasone to the local anesthetic. Blinding the performer will help to eliminate performance bias. Two 20 cc syringes of 0.5% ropivacaine will be prepared for the block. One cc of the study drug will be injected into each syringe and mixed.

Before nerve blockade, all patients will receive intravenous access and standard monitoring, which included noninvasive blood pressure, electrocardiogram, and pulse oximetry.

Sedation and anxiolysis are achieved with intravenously administered midazolam in 1- to 2-mg increments up to 5 mg and fentanyl in 25 ug increments as needed up to 250 ug.

POPLITEAL NERVE BLOCK

Popliteal nerve block will be performed with the patient lying supine and the operative leg propped up on an elevation pillow allowing the posterior popliteal fossa to be accessed. A linear, high-frequency US probe of 5 to 12 MHz (S-nerve, sonosite) covered with a sterile dressing will be placed in the popliteal fossa in a transverse plane. The tibial and common peroneal nerve are identified superficial and lateral to the popliteal vessels then traced cephalad until they unite. This is the point of needle placement.

After sterilization and application of LA (3ml of 0.5% lidocaine) to the skin, a 22-gauge, Tuohy is advanced through the skin at the lateral border thigh in alignment with the long axis of the ultrasound probe in the same plane as the US beam (ie, in-plane technique). The needle is to be positioned under US guidance to the tibial nerve and common peroneal nerve.

The needle is to be always visualized before LA injection. Hydrolocation or dissection beyond 3 cc is not to be used to avoid dilution effect. Once needle position was satisfactory and after negative aspiration, 10 mL of LA is to be injected incrementally over 2 minutes with direct sonographic visualization of the LA spread around the tibial nerve. The needle is to be repositioned under US guidance to ensure adequate spread of LA around the tibial nerve. A circumferential spread of the LA is sought. Extra care is taken never to inject within the nerve. Expansion and compartmentalization of the nerve structure will result in abandonment of the study. Similarly, 10 ml of LA is injected circumferentially around the common peroneal nerve.

FEMORAL NERVE BLOCK

1. A femoral nerve block is placed in the usual manner of our institutional practice. Femoral nerve block will be performed with the patient lying supine. A linear, high-frequency US probe of 5 to 12 MHz (S-nerve, sonosite) covered with a sterile dressing will be placed on the inguinal crease in a transverse plane. The femoral artery is identified and traced cephalad until the profundus branch joins the femoral artery proper. This is the level of needle placement.
2. After sterilization and application of LA (3ml of 1% lidocaine) to the skin, a 19-gauge, Tuohy is advanced through the skin at the lateral border of the upper thigh in alignment with the long axis of the ultrasound probe in the same plane as the US beam (ie, in-plane technique). The needle is to be positioned under US guidance to the lateral and anterior portion of the femoral nerve.
3. The needle is to be always visualized before LA injection. No more than 3cc of hydrolocation or hydrodissection is allowed. Once needle position was satisfactory and after negative aspiration, a 20 mL syringe containing 20 mL of LA where 10mL is to be injected incrementally over 3 minutes with direct sonographic visualization of the LA spread. The needle is to be repositioned under the femoral nerve US guidance to ensure adequate spread of LA above the nerves using the remaining 5 mL of LA. A circumferential spread of the LA is sought. Extra care is taken never to inject within the nerve.

OBTURATOR NERVE BLOCK The single shot obturator nerve block is performed with the patient lying supine with the leg slightly abducted and flexed at the hip joint. The same ultrasound probe is used and positioned more medially to locate the fascial plane between the adductor brevis and adductor magnus where the posterior division of the obturator nerve lies. After local infiltration of the skin with 3cc of 1% lidocaine, a 22 G Tuohy needle is advanced in plane with until it lies within the fascial plane of the adductor magnus and adductor brevis. No more than 3 cc of hydrolocation or hydrodissection is allowed. 5 cc of ropivacaine is injected here taking care that hydrodissection of the fascial plane occurs and avoiding intramuscular injection.

INTRAOP General anesthesia is performed in the usual fashion. Fentanyl is used intraoperatively if the heart rate or blood pressure deviated greater than 20% from the baseline if deemed appropriate. No other opioid or analgesics (such as ketorolac or ketamine) will be given as per institutional practice. If there is suspicion that the blocks are not working intraoperatively, the patient may be withdrawn from the study and alternative analgesia may be given. The dexamethasone or sham is given at the beginning of the surgery and ondansetron 4 mg is given at the end of surgery.

POST-ANESTHESIA CARE UNIT In PACU, the patient is evaluated for femoral, sciatic and obturator block success. If any of the 3 blocks are deemed non functional, the patient is withdrawn from the study and noted.

The patient will be given hydromorphone 0.2mg IV boluses in PACU to maintain the VAS score below 4 if necessary. The standard institutional hydromorphone PCA set at 0.2mg bolus every 10 minutes with no basal.

At the time of discharge from PACU, the patients are given a diary to record their perception of sensation and movement every awake hour on a scale of 0 to 2. Zero being no sensation, 1 = some sensation and 2 being full sensation being recorded separately on top of the foot and on the bottom of the foot. Similarly a 0 to 2 scale for strength. 0 being no movement, 1= some movement, 2 = full strength in pointing the toes towards the nose and in pointing the toes away from the nose.

Patients will also be given instructions to record the location of their pain when it first returns and each time they require pain medications; being on top or at the bottom of the knee.

FOLLOW UP All patients will be be seen the day after the surgery for their time to first return of sensation and time to first return of movement. Also information regarding the full return of sensation and time to full return of movement is obtained. If sensory and motor function remains intact, a further interview will be conducted daily until full sensory and motor function returns. All complications will be noted.

All patients will have their PCA and medication records checked for the time of their first request for analgesia. Patients will be interviewed on the location of their pain for this request for analgesia if the patient's pain location record is ambiguous.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I to III,
* Aged 18 and above,
* Undergoing total knee replacement.

Exclusion Criteria:

* Body mass index of more than 45 kg/m2 (higher chance of failure)
* Weight less than 70 kg
* Diabetes
* Injection site deformities
* Infection at the injection site
* Existing peripheral neuropathy
* Allergy to LA agents
* Contraindications to dexamethasone
* Patients with severe PONV
* Patients with peptic ulceration or upper GI bleed of unknown origin
* Coagulopathy
* Any other contraindication to lower limb peripheral nerve block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Duration of Analgesia | 72 hours or first report of pain in the knee which ever is earliest
  Duration of analgesia defined as the time interval between the end of local anesthetic injection and the patient's first report of pain in the knee.

SECONDARY OUTCOMES:
Duration of motor blockade | 72 hour or first return of motor function
  Time interval between the end of local anesthetic injection and the patient's first report of return in motor function in femoral, obturator and sciatic distribution
Duration of sensory blockade | 72 hours or first report of sensory recovery
  Time interval between the end of local anesthetic injection and the patient's first report of return in any sensation in the distribution of femoral and sciatic distribution
Complete sensory return | 72 hours or when the patient first reports complete sensation
  interval between the end of local anesthetic injection and the patient's first report of return in complete sensation in the distribution of femoral and sciatic distribution

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Lam, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States